CLINICAL TRIAL: NCT04951050
Title: A Prospective, Multicenter, Single-arm Trail in Evaluating the Safety and Efficacy of the Rapamycin Target Eluting Stent in Patients With Coronary Artery Stenosis
Brief Title: TARGET-PREMIER Trail in Evaluating the Safety and Efficacy of the Rapamycin Target Eluting Stent in CAS Treatment
Acronym: T-P
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-IC-035
Record Dates: First submitted 2021-06-26; First posted 2021-07-06 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Coronary Stenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug eluting stent (Experimental)
  Interventions: Device: Rapamycin target eluting stent

INTERVENTIONS:
Device: Rapamycin target eluting stent — Rapamycin target eluting stent

SUMMARY:
The aim of the TARGET PREMIER trail in to demonstrate the safety and efficacy of the rapamycin target eluting stent in the treatment of subjects with ischemic heart disease (asymptomatic myocardial ischemia , table or unstable angina), with target lesion(s) in coronary arteries with visually estimated reference vessel diameter ≥2.25mm and ≤4.0 mm.

DETAILED DESCRIPTION:
200 participants with coronary artery stenosis will enrolled in the investigation to receive PCI surgery treatment with rapamycin target eluting stent implantation. All the participants will get clinical follow-up after PCI surgery within 30 days, 6 months, 9 months, 12 months and 2-5 years, and they will be conducted coronary angiogram at 9th month after PCI to get the data of in-stent late loss which was the main endpoint of the investigation. The secondary endpoints including device sucess, operation success, clinical sucess, Doce, PoCE, TLR, TVR, MI incident rate, death, stent thrombosis as defined by ARC, stent retraction, MLD, DS and ARB. The data derived from the investigation will be performed statistic analysis to evaluate whether the clinical outcome meet the PG.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patient with an indication for percutaneous coronary intervention (PCI) including silent ischemia (in absence of symptoms a positive functional study or a reversible change in the ECG consistent with ischemia), angina (stable or unstable).
3. Subject acceptable candidate for coronary artery bypass surgery (CABG).
4. Patient or legal guardian is willing and able to provide informed written consent and comply with follow-up visits and testing schedule.

Angiographic Inclusion Criteria:

1. Treatment up to two target lesions with a maximum of two lesions per epicardial vessel. If there are two target lesions within the same epicardial vessel, the two target lesions must be at least 10mm apart per visual estimation.
2. Target lesion(s) must be located in a native coronary artery with a visually estimated diameter stenosis ≥70%, TIMI 1, lesions length ≤36mm. Target vessel must be visually estimated diameter of ≥2.25mm to ≤4.0mm.
3. Target lesion must be adequately covered with a single stent.
4. Up to two target lesion needed treatment in one target vessel.
5. One non-target lesion is allowed prior to enrollment if successful. It should be located at the distal end of the target lesion, and be at lease 10mm apart, when both are in the same epicardial vessel.

Exclusion Criteria:

General Exclusion Criteria:

1. Acute myocardial infarction with 1 week or enzyme levels (Creatinkinase or Troponin) demonstrating that either or both enzyme levels have not returned to normal limits at the time of the procedure.
2. Target vessel (including branches) PCI within 12 months of the baseline procedure.
3. Known congestive heart failure (NYHA III) or left ventricular ejection fraction (LVEF) <30%
4. Patient has current unstable arrhythmias.
5. Patient has a history of any coronary arteries brachytherapy.
6. Planned surgery within 6 months after index procedure.
7. Platelet count <100,000 cells/mm3 or >700,000 cells/mm3, white blood cell (WBC) count <3,000 cells/mm3.
8. Impaired renal function (serum creatinine >2.0mg/dl) or patient on dialysis.
9. Cerebrovascular accident or transient ischemic attack within the past 6 months, or any permanent neurologic defect attribute to cerebral vascular accident (CVA).
10. Patient has a history of bleeding diathesis, contraindication to dual antiplatelet therapy (DAPT).
11. Known allergy to protocol-required concomitant medications such as aspirin, or clopidogrel, or heparin and the study stent components such as cobalt, nickel, chromium, rapamycin or similar drugs.
12. Patient is participating in or plans to participate in any other investigational drug or device clinical trial that has not reached its primary endpoint.
13. Other serious medical illness with life expectancy less than 1 year (e.g. cancer, congestive heart failure).
14. Patient has immunosuppressive or autoimmune disease, and is receiving or scheduled to immunosuppressive therapy.
15. A
16. Women who are pregnant or breastfeeding (women of child-bearing potential must have a negative pregnancy test with on week before treatment.)
17. Women who intend to become pregnant with 12 months after the baseline procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the baseline procedure).
18. Patient has received an organ transplant or is on a waiting list for an organ transplant.
19. Patient is receiving or scheduled to receive chemotherapy or radiotherapy with 30 days before or any time after the baseline procedure.
20. Patient may not be obedient to the clinical investigation plan through the judgment by investigators.

Angiographic Inclusion Criteria:

1. Left main artery coronary disease.
2. Three-vessel coronary artery disease.
3. Target lesion is located in or supplied by an arterial or venous bypass graft.
4. In-stent restenosis lesions.
5. Patient has additional lesion(s) for which an intervention with 1 year after the index procedure would be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-08-26 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
In-stent late loss | 9 months
  In-stent late loss at 9 months post-procedure as measured by quantitative coronary angiography (QCA)

SECONDARY OUTCOMES:
Target Lesion Failure | 30days, 6 months, 9months, 12 months and yearly thereafter until 5 years
  Percentage of participants that had either Cardiac Death, Myocardial Infarction (not clearly attributable to a non-target vessel)or Target Lesion Revascularization (TLR, clinically indicated)
Any myocardial ischemia (MI) | 30days, 6 months, 9months, 12 months and yearly thereafter until 5 years
  percentage of participants that had any MI
Any revascularization | 30days, 6 months, 9months, 12 months and yearly thereafter until 5 years
  percentage of participants that had any revascularization
Ischemia-driven TLR | 30days, 6 months, 9months, 12 months and yearly thereafter until 5 years
  percentage of participants that had Ischemia-driven TLR
Probable and definite stent thrombosis defined by Academic Research Consortium (ARC) | 30days, 6 months, 9months, 12 months and yearly thereafter until 5 years
  percentage of participants that had probable and definite stent thrombosis
Late lumen loss in segment | 9 months
  Late Lumen Loss in segment at 9 months post-procedure as measured by quantitative coronary angiography (QCA)
In-stent and in-segment binary restenosis rate | 9 months
  percentage of restenosis ≥50% in-stent or in-segment at 9 months post-procedure
Device success | 0 day
  Device Success is defined as a final residual diameter stenosis of <30%, thrombolysis in myocardial infarction (TIMI) 3, by QCA, using the assigned device only
Procedure success | During the hospital stay to a maximum of the first seven days post index procedure
  Procedure Success defined as achievement of a final diameter stenosis of <30%, TIMI 3, by QCA, using any percutaneous method, without the occurrence of death, Q-wave or non-Q-wave MI, or repeat revascularization of the target lesion during the hospital stay.
Target lesion success | 0 day
  Target lesion success defined as achievement of a final diameter stenosis of <30%, TIMI 3, by QCA, using any percutaneous method.
TLR | 30days, 6 months, 9months, 12 months and yearly thereafter until 5 years
  Including ischemia driven or non-ischemia driven
target vessel revascularization (TVR) | 30days, 6 months, 9months, 12 months and yearly thereafter until 5 years
  Including ischemia driven or non-ischemia driven
Patient oriented composite endpoint (PoCE) | 30days, 6 months, 9months, 12 months and yearly thereafter until 5 years
  defined as all death, all MI and any revascularization
In-stent and in-segment %diameter stenosis (%DS) | 9 months
  In-stent and in-segment %diameter stenosis (%DS) at 9 months post-procedure as measured by QCA
In-stent and in-segment minimum lumen diameter | 9 months
  In-stent and in-segment minimum lumen diameter at 9 months post-procedure as measured by QCA.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Xiong Zhong, MD, Principal Investigator — Meizhou Peple's Hospital in Guangdong Province
Locations (1):
- Meizhou Peple's Hospital, Meizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No